CLINICAL TRIAL: NCT01801566
Title: Effectiveness of the Single Implant-retained Mandibular Overdenture Treatment: Radiographic Evaluations, Patient's Satisfaction, and Oral-health-related Quality of Life
Brief Title: Effectiveness of the Single Implant-retained Mandibular Overdenture Treatment
Acronym: SIOver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Associate professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1129-9956
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Mouth, Edentulous
Keywords: Mandibular Prosthesis Implantation; Prostheses and Implants; Denture, Complete, Lower
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional implant loading protocol (Active Comparator): Single implant-retained mandibular overdenture
  Interventions: Procedure: Single implant-retained mandibular overdenture
- Immediate loading implant protocol (Experimental): Single implant-retained mandibular overdenture
  Interventions: Procedure: Single implant-retained mandibular overdenture

INTERVENTIONS:
Procedure: Single implant-retained mandibular overdenture — 60 patients treated with single implant retained complete mandibular denture (overdenture) opposed to a conventional maxillary denture, allocated into 2 experimental groups according to the implant loading protocol (conventional and immediate), evaluated at baseline and after 1, 3, 6 and 12 months after treatment.

SUMMARY:
This study aims to evaluate the treatment with single implant overdenture for the edentulous mandible. The investigators hypothesize that treatment with lower overdenture retained by a single implant appears to have satisfactory effectiveness as a treatment for patients with specific conditions (such as maladaptive patients), with the advantages of simplicity and greater immediate benefits when compared to the conventional full denture, improving the retention and stability of the denture and better oral-related quality of life.

DETAILED DESCRIPTION:
This study is a longitudinal evaluation of clinical and patient-reported outcomes related to the single-implant mandibular overdenture treatment. Sixty completely edentulous individuals will be included. First, new complete dentures will be fabricated for all of them. Panoramic radiographs and conventional tomograms of the mandibular midline region will be obtained in order to plan the implant placement surgery. After the adaptation period related to the use of the new dentures, a single implant (Titamax IT Cortical, Neodent, Curitiba, Brazil) will be installed in the mandibular midline of all participants. According to the primary stability obtained in the implant placement patients will be treated with an immediate loading protocol when achieving torque of at least 30 Ncm and implant stability quotient (ISQ) of at least 60. In cases of values below cited, conventional loading protocol will be adopted. Ball O-ring will be used as the attachment system for the mandibular overdenture. Clinical and patient-reported outcomes will be collected after 1, 3, 6 and 12 months after the installation of the overdentures.

ELIGIBILITY:
Inclusion Criteria:

* Fully edentulous patients
* Need of replacement of the mandibular denture or patient without mandibular denture
* Patients with poor adaptation to the mandibular denture
* Patients with good general health

Exclusion Criteria:

* Patients who refuse to receive a conventional dentures opposed to a mandibular overdenture retained by a single implant
* Patients with local intraoral diseases that influence denture stability, retention and adaptation of the lower denture (such as changes or anatomical deformations of the jaws, mucosal changes caused by fungi and bacteria, tumor changes and absolute xerostomia)
* Patients with systemic, psychological or neurological diseases that preclude or hinder oral movements of the patient for clinical care and/or clinical follow-up in all stages of the research
* Patients who choose other treatment modalities not covered by the study
* Patients with alcoholism or other severe behavioral disorders that compromise their participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life impacts | Change from baseline on oral health-related quality of life impacts at 12 months
  Oral health related quality of life impacts were measured using the Brazilian version of the Oral Health Impact Profile for Edentulous subjects (Souza et al., 2007; Souza et al., 2010), considering the overall scale and its four different scale domains: masticatory discomfort and disability (four items), (2) psychological discomfort and disability (five items), social disability (five items) and oral pain and discomfort (five items).

SECONDARY OUTCOMES:
Satisfaction with dentures | Change from baseline on satisfaction with dentures at 12 months
  Satisfaction with dentures measured using the patients' ratings of the overall satisfaction with the mandibular denture, and satisfaction with comfort, stability, esthetics, ability to speak, and ability to chew. All satisfaction items will be measured on a 10-point visual analogue scale ranging from 0 to 10

OTHER OUTCOMES:
Primary stability | Changes from baseline on primary stability of implants at 12 months
  Measures of the implant stability: stability quotient index and final insertion torque
Crestal bone loss | Changes from baseline on crestal bone loss at 12 months
  Periimplant alveolar bone height of the crestal bone level
Bone density around the implant | Changes from baseline on bone density around the implant at 12 months
  Periimplant bone density measured by digital subtraction radiography

CONTACTS AND LOCATIONS:
Overall Officials: Claudio R Leles, DDS, PhD, Principal Investigator — Universidade Federal de Goias
Locations (1):
- School of Dentistry, Federal University of Goias, Goiânia, Goiás, Brazil

REFERENCES:
- See also: Website of the Main study sponsor — http://cnpq.br/